CLINICAL TRIAL: NCT01656278
Title: Does an MRI-guided Treatment Strategy Reduce Disease Activity and Progression in Patients With Rheumatoid Arthritis (RA): a Randomised Controlled Trial
Brief Title: An MRI-guided Treatment Strategy to Prevent Disease Progression in Patients With Rheumatoid Arthritis
Acronym: IMAGINE-RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor of Rheumatology, MD, DMSci, Kim Horslev-Petersen (Other)
Collaborators: King Christian X´Hospital for Rheumatic Diseases (Other); Slagelse Hospital (Other); Glostrup University Hospital, Copenhagen (Other); Abbott (Industry)
Responsible Party: Sponsor-Investigator, Professor of Rheumatology, MD, DMSci, Kim Horslev-Petersen, Professor of Rheumatology, MD, DMSci, King Christian X´Hospital for Rheumatic Diseases
Organization: King Christian X´Hospital for Rheumatic Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMAGINE-RA
Record Dates: First submitted 2012-07-05; First posted 2012-08-02 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Arthritis; Arthritis, Rheumatoid; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Connective Tissue Diseases; Autoimmune Diseases
Keywords: Arthritis, Rheumatoid/drug therapy; Arthritis, Rheumatoid/pathology; Disease Progression; Longitudinal Studies; Prospective Studies; Imaging, Magnetic Resonance; Remission Induction; Synovitis/immunology; Synovitis/pathology; Wrist Joint/pathology; Wrist Joint/physiopathology
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Connective Tissue Diseases; Autoimmune Diseases; Disease Progression; Synovitis | interventions — Magnetic Resonance Spectroscopy; Restraint, Physical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional biochemical and clinical examinations (Active Comparator): Biochemical and clinical examinations
  Interventions: Other: Conventional biochemical and clinical examinations
- Conventional biochemical and clinical examinations and MRI. (Experimental): Biochemical and clinical examinations and MRI.
  Interventions: Procedure: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Procedure: Magnetic resonance imaging (MRI) — Treatment algorithm based on conventional biochemical/clinical examinations AND MRI of unilateral 2nd to 5th MCP joints and wrist on dominant side. Assessed month 0, 4, 8, 12, 16, 20, 24 with treatment intensification after predefined treatment algorithm in the case of "unsatisfactory inflammatory activity", which is defined as the presence of at least one physically swollen joint and DAS28>3.2 AND/OR MRI-detected bone marrow oedema score > 0 (RAMRIS-score)
  Arms: Conventional biochemical and clinical examinations and MRI.
Other: Conventional biochemical and clinical examinations — Treatment algorithm based on conventional biochemical and clinical examinations. Assessed month 0, 4, 8, 12, 16, 20, 24 with treatment intensification after predefined treatment algorithm in the case of "unsatisfactory inflammatory activity", which is defined as the presence of at least one clinically swollen joint and DAS28>3.2
  Arms: Conventional biochemical and clinical examinations

SUMMARY:
The purpose of this study is to examine whether an magnetic resonance imaging (MRI) -guided treatment strategy based on a predefined treatment algorithm can prevent progression of erosive joint damage, increase remission rate and improve functional level in the short and long term in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory joint disease. Patients typically experience pain, functional impairment and reduced quality of life, and are at risk of developing progressive joint damage. The disease primarily affects the small joints of the hands and feet. The current treatment strategy involves early and intensive treatment with close clinical follow up, which attempts to control the disease and avoid inflammation and thereby prevent pain, improve functional level and avoid joint damage. It is therefore important for optimal treatment of RA patients that methods used for diagnosis, disease monitoring and prognostication are highly sensitive. Erosive joint damage occurs early in the disease. Joint deformity is irreversible and causes serious functional impairment. Early and intensive treatment with close monitoring of the inflammation can slow the destructive disease and prevent function loss. However, it has been demonstrated that patients who are shown by conventional clinical and biochemical examination to have low disease activity or to be in remission can still have progressive joint damage. This demonstrates that current clinical/biochemical methods used in daily clinical practice are not sufficiently sensitive and other methods are required for the monitoring of disease activity and prognostication.

The presence of erosions (shown by X-ray examination) as well as anti-cyclic citrullinated peptide (anti-CCP) antibodies and bone marrow oedema (osteitis) on magnetic resonance imaging (MRI), are all independent predictors of subsequent radiographic progression. Bone marrow oedema has been shown to be the strongest independent predictor in early RA and MRI therefore has significant prognostic value.

It is therefore possible that supplementing conventional clinical and biochemical examinations of RA patients with MRI, and intensifying treatment where bone marrow oedema is present, will help reduce disease activity, avoid progressive joint damage and prevent function loss.

The current study is therefore based on the following hypothesis:

By supplementing conventional clinical and biochemical examination of RA patients with low disease activity/in remission with MRI and intensifying treatment in the case of sub-clinical inflammation as measured by the presence of bone marrow oedema, it is possible to prevent radiographic erosive progression, improve functional level and enable more patients to achieve clinical remission.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* RA according to ACR (American College of Rheumatology)/EULAR (European League Against Rheumatism) 2010 criteria.
* Anti-CCP positivity
* Erosions on conventional X-ray of hands, wrists and/or feet
* No clinically swollen joints
* DAS28 (4 variable, CRP) < 3.2
* DMARD monotherapy treatment OR combination treatment, in the form of 2- or 3-drug therapy. If the patient is undergoing 3-drug therapy, at least one of the preparations must be administered at less than the "maximum inclusion dose"*
* Unchanged anti-rheumatic treatment in the previous 6 weeks or more
* No previous treatment with biological medication
* No contra-indications for TNF-alpha-inhibiting treatment
* No contra-indications for MRI
* s-creatinine within normal range
* Ability and willingness to give written and oral informed consent and fulfil the requirements of the study programme with reference to the protocol

  * Maximum "inclusion dose" is defined as: MTX 25 mg/week (or maximum tolerated dose if 25 mg/week is not tolerated), SSZ 2g/day (or maximum tolerated dose if 2 g/day is not tolerated) and HCQ 200 mg/day (or maximum tolerated dose if 200 mg/day is not tolerated)

Exclusion Criteria:

* Previous or current biological treatment
* Known intolerance to methotrexate treatment which means that the patient is not able to tolerate a minimum of MTX 7.5 mg (minimum dose).
* DMARD 3-drug therapy at maximum tolerated/maximum "inclusion dose"*
* I.m, intra-articular or i.v glucocorticoid administration ≤ 6 weeks prior to inclusion
* Oral glucocorticoid administration > 5 mg/day
* Changes in oral glucocorticoid dose < 3 months prior to inclusion
* Myocrisin treatment
* Affected liver enzymes > 2 x the upper limit of normal at the time of screening
* Current and/or imminent wish to become pregnant
* Contra-indications for TNF-alpha-inhibiting treatment
* Contra-indications for MRI
* Known alcohol/drug abuse
* Inability to give informed consent
* Inability to cooperate with the study programme due to physical or mental reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
DAS28 remission (<2.6) | 24 month
No radiographic progression (assessed by the Sharp/vdHeijde method). | 24 month

SECONDARY OUTCOMES:
No radiographic progression (Sharp/vdHeijde score). | 24 month
  No radiographic progression (Sharp/vdHeijde score) from 0-12 and 12-24 months and change in Sharp/vdHeijde score from 0-12, 0-24 and 12-24 months.
No MRI erosion (RAMRIS) score | 24 month
  No progression in MRI erosion (RAMRIS) score from 0-12 and 12-24 months and change in MRI erosion (RAMRIS) score from 0-12, 0-24 and 12-24 months.
MRI synovitis (RAMRIS) score | 24 months
  MRI synovitis (RAMRIS) score at 12 and 24 months
MRI bone marrow oedema (RAMRIS) score | 24 months
  MRI bone marrow oedema (RAMRIS) score at 12 and 24 months
HAQ score | 24 month
  Changes in HAQ score from 0-12 and 0-24 months
SF-36 score | 24 month
  Changes in SF-36 score from 0-12 and 0-24 months
EQ-5D score | 24 month
  Changes in EQ-5D score from 0-12 and 0-24 months
ACR/EULAR 2011 remission | 24 month
  ACR/EULAR 2011 remission at 12 and 24 months
DAS28 | 24 month
  DAS28 at 12 and 24 month
DAS28 remission (<2.6) at 12 months | 24 months
biomarker analyses | 24 month

OTHER OUTCOMES:
Dynamic MRI | 24 month
  Dynamic MRI variable (including initial rate of enhancement (IRE) and maximum enhancement (ME)).

CONTACTS AND LOCATIONS:
Overall Officials: Kim Hørslev-Petersen, Professor, Principal Investigator — King Christian X´Hospital for Rheumatic Diseases; Signe Møller-Bisgaard, MD, Study Director — Dep. of Rheumatology, Rigshospitalet, Glostrup; Mikkel Østergaard, Professor, Study Chair — Dep. of Rheumatology, Rigshospitalet, Glostrup; Bo Ejbjerg, MD, PhD, Study Chair — Dep. of Rheumatology Slagelse Hospital; Merete Hetland, MD, PhD, DMSci, Study Chair — Dep. of Rheumatology, Rigshospitalet, Glostrup
Locations (9):
- Denmark (9):
  - Dep. of Rheumatology Aarhus Hospital, Aarhus
  - Dep. of Rheumatology Frederiksberg Hospital, Copenhagen
  - Dep. of Rheumatology Glostrup Hospital, Copenhagen
  - Dep. of Rheumatology Gentofte Hospital, Copenhagen
  - Dep. of Rheumatology King Christian X´Hospital for Rheumatic Diseases, Gråsten
  - Department of Rheumatology University Hospital Vendsyssel, Hjørring
  - Dep. of rheumatology Odense Hospital, Odense
  - Dep. of Rheumatology Silkeborg Hospital, Silkeborg
  - Dep. of Rheumatology Slagelse Hospital, Slagelse

REFERENCES:
- [Derived] Moller-Bisgaard S, Horslev-Petersen K, Ejbjerg B, Hetland ML, Christensen R, Ornbjerg LM, Glinatsi D, Moller JM, Boesen M, Stengaard-Pedersen K, Madsen OR, Jensen B, Villadsen JA, Hauge EM, Bennett P, Hendricks O, Asmussen K, Kowalski M, Lindegaard H, Bliddal H, Krogh NS, Ellingsen T, Nielsen AH, Larsen L, Jurik AG, Thomsen HS, Ostergaard M. Effect of initiating biologics compared to intensifying conventional DMARDs on clinical and MRI outcomes in established rheumatoid arthritis patients in clinical remission: Secondary analyses of the IMAGINE-RA trial. Scand J Rheumatol. 2022 Jul;51(4):268-278. doi: 10.1080/03009742.2021.1935312. Epub 2021 Sep 2. PMID 34474649
- [Derived] Moller-Bisgaard S, Georgiadis S, Horslev-Petersen K, Ejbjerg B, Hetland ML, Ornbjerg LM, Glinatsi D, Moller J, Boesen M, Stengaard-Pedersen K, Madsen OR, Jensen B, Villadsen JA, Hauge EM, Bennett P, Hendricks O, Asmussen K, Kowalski M, Lindegaard H, Bliddal H, Krogh NS, Ellingsen T, Nielsen AH, Balding L, Jurik AG, Thomsen HS, Ostergaard M. Predictors of joint damage progression and stringent remission in patients with established rheumatoid arthritis in clinical remission. Rheumatology (Oxford). 2021 Jan 5;60(1):380-391. doi: 10.1093/rheumatology/keaa496. PMID 32929463
- [Derived] Moller-Bisgaard S, Horslev-Petersen K, Ejbjerg B, Hetland ML, Ornbjerg LM, Glinatsi D, Moller J, Boesen M, Christensen R, Stengaard-Pedersen K, Madsen OR, Jensen B, Villadsen JA, Hauge EM, Bennett P, Hendricks O, Asmussen K, Kowalski M, Lindegaard H, Nielsen SM, Bliddal H, Krogh NS, Ellingsen T, Nielsen AH, Balding L, Jurik AG, Thomsen HS, Ostergaard M. Effect of Magnetic Resonance Imaging vs Conventional Treat-to-Target Strategies on Disease Activity Remission and Radiographic Progression in Rheumatoid Arthritis: The IMAGINE-RA Randomized Clinical Trial. JAMA. 2019 Feb 5;321(5):461-472. doi: 10.1001/jama.2018.21362. PMID 30721294
- [Derived] Moller-Bisgaard S, Horslev-Petersen K, Ejbjerg BJ, Boesen M, Hetland ML, Christensen R, Moller J, Krogh NS, Stengaard-Pedersen K, Ostergaard M. Impact of a magnetic resonance imaging-guided treat-to-target strategy on disease activity and progression in patients with rheumatoid arthritis (the IMAGINE-RA trial): study protocol for a randomized controlled trial. Trials. 2015 Apr 21;16:178. doi: 10.1186/s13063-015-0693-2. PMID 25896862